CLINICAL TRIAL: NCT00553098
Title: Hematopoietic Cell Transplantation for Treatment of Patients With Primary Immunodeficiencies and Other Nonmalignant Inherited Disorders Using Low-Dose TBI and Fludarabine With or Without Campath®
Brief Title: Alemtuzumab, Fludarabine Phosphate, and Total-Body Irradiation Followed by a Donor Stem Cell Transplant in Treating Patients With Immunodeficiency or Other Nonmalignant Inherited Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Lauri Burroughs, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007.00; NCI-2009-01550 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2007; 2007.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Immunodeficiency Syndrome; Non-Cancer Diagnosis
MeSH Terms: conditions — Immunologic Deficiency Syndromes | interventions — Alemtuzumab; Cyclosporine; Cyclosporins; fludarabine phosphate; Mycophenolic Acid; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (chemotherapy, low dose radiation) (Experimental): CONDITIONING REGIMEN: *Patients with no life-threatening viral or fungal infections within 1 month before the planned HCT receive alemtuzumab IV over 6 hours on day -10 and fludarabine phosphate IV over 30 minutes on days -4 to -2. They also undergo low-dose TBI on day 0. Patients with HLH, IPEX syndrome, DiGeorge syndrome, or life-threatening viral or fungal infections within 1 month before the planned HCT receive fludarabine phosphate IV over 30 minutes on days -4 to -2 and undergo 2 low doses of TBI on day 0.
  HEMATOPOIETIC CELL TRANSPLANTATION: Patients undergo HCT on day 0.
  IMMUNOSUPPRESSION: Patients receive cyclosporine IV or PO 2-3 times daily beginning on day -3 and continuing until day 100 followed by a taper until day 180. They also receive mycophenolate mofetil IV or PO 3 times daily beginning on day 0 and continuing until day 40 followed by a taper until day 96.
  Interventions: Biological: Alemtuzumab; Procedure: Allogeneic Bone Marrow Transplantation; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Cyclosporine; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Radiation: Total-Body Irradiation

INTERVENTIONS:
Biological: Alemtuzumab — Given IV
  Other Names: Anti-CD52 Monoclonal Antibody; Campath; Campath-1H; LDP-03; MabCampath; Monoclonal Antibody Campath-1H
Procedure: Allogeneic Bone Marrow Transplantation — Undergo HCT
  Other Names: Allo BMT; Allogeneic BMT
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo HCT
  Other Names: allogeneic stem cell transplantation; HSC; HSCT
Drug: Cyclosporine — Given PO or IV
  Other Names: 27-400; Ciclosporin; CsA; Cyclosporin; Cyclosporin A; Neoral; OL 27-400; Sandimmun; Sandimmune; SangCya
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; Oforta; SH T 586
Other: Laboratory Biomarker Analysis — Correlative study
Drug: Mycophenolate Mofetil — Given PO or IV
  Other Names: Cellcept; MMF
Radiation: Total-Body Irradiation — Undergo low dose TBI
  Other Names: TOTAL BODY IRRADIATION; Whole-Body Irradiation

SUMMARY:
This phase II trial studies fludarabine phosphate and total-body irradiation with or without alemtuzumab followed by donor stem cell transplant to see how well it works in treating patients with immunodeficiency or other nonmalignant inherited disorders. Giving chemotherapy, such as fludarabine phosphate, a monoclonal antibody such as alemtuzumab, and radiation therapy before a donor stem cell transplant helps stop the growth of abnormal cells. It may also stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining abnormal cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Improve donor chimerism levels in patients with inherited nonmalignant disorders undergoing hematopoietic cell transplantation (HCT) using a reduced intensity conditioning regimen either through the addition of Campath (alemtuzumab) or a slightly higher dose of total-body irradiation (TBI).

SECONDARY OBJECTIVES:

I. Decrease the incidence and severity of acute and chronic graft-versus-host disease (GVHD) through use of marrow as the stem cell source and Campath.

II. Assess disease response following HCT.

III. Immune reconstitution following HCT.

IV. Incidence of infections.

V. Overall survival.

VI. Percent of patients with cluster of differentiation (CD)33/CD19 donor chimerism > 50%.

OUTLINE:

CONDITIONING REGIMEN: Patients with no life-threatening viral or fungal infections within 1 month before the planned hematopoietic cell transplantation (HCT) receive alemtuzumab intravenously (IV) over 6 hours on day -10 and fludarabine phosphate IV over 30 minutes on days -4 to -2. They also undergo low-dose TBI on day 0. Patients with hemophagocytic lymphohistiocytosis (HLH), immune dysregulation polyendocrinopathy enteropathy X-linked (IPEX) syndrome, DiGeorge syndrome, or life-threatening viral or fungal infections within 1 month before the planned HCT receive fludarabine phosphate IV over 30 minutes on days -4 to -2 and undergo 2 low doses of TBI on day 0.

HEMATOPOIETIC CELL TRANSPLANTATION: Patients undergo HCT on day 0.

IMMUNOSUPPRESSION: Patients receive cyclosporine IV or orally (PO) 2-3 times daily beginning on day -3 and continuing until day 100 followed by a taper until day 180. They also receive mycophenolate mofetil IV or PO 3 times daily beginning on day 0 and continuing until day 40 followed by a taper until day 96.

After completion of HCT, patients are followed up at day 84, at 6, 12, 18 and 24 months post-transplantation, and then once a year for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Primary immunodeficiency disorder or other nonmalignant inherited disease (except aplastic anemia and Fanconi anemia) treatable by allogeneic HCT
* Patients with pre-existing medical conditions or other factors that renders them at high risk for regimen related toxicity or ineligible for a conventional myeloablative HCT
* Donors: Related donor who is human leukocyte antigen (HLA) genotypically identical at least at one haplotype and may be genotypically or phenotypically identical for serological typing for HLA-A, B, -C, and at the allele level for -DRB1 and -DQB1; related donors must be a match or a single allele mismatch at HLA-A, B, and C (at highest resolution available at the time of donor selection) and matched at DRB1 and DQB1 by deoxyribonucleic acid (DNA) typing
* Donors: Unrelated donors who are prospectively:

  * Matched for HLA-A, B, C, DRB1 and DQB1 by DNA typing at the highest resolution routinely available at the time of donor selection
  * Only a single allele disparity will be allowed for HLA-A, B, or C as defined by high resolution typing (no mismatching for DRB1 or DQB1 is allowed)

Exclusion Criteria:

* Patients with Aplastic anemia and Fanconi anemia
* Patients with metabolic storage diseases who have severe central nervous system (CNS) involvement of disease, defined as intelligence quotient (IQ) score < 70
* Cardiac ejection fraction < 30% or, if unable to obtain ejection fraction, shortening fraction of < 26%) on multi-gated acquisition (MUGA) scan or cardiac echo, symptomatic coronary artery disease, other cardiac failure requiring therapy; patients with a history of, or current cardiac disease should be evaluated with appropriate cardiac studies and/or cardiology consult; patients with a shortening fraction < 26% may be enrolled if approved by a cardiologist
* Poorly controlled hypertension despite anti-hypertensive medications
* Patients with clinical or laboratory evidence of liver disease will need to be evaluated for the cause of the liver disease, its clinical severity in terms of liver function and the degree of portal hypertension; patients will be excluded if they are found to have: fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, bridging fibrosis, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evidenced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3mg/dl, or symptomatic biliary disease (Patients will be allowed on to the protocol with liver problems if gastroenterology approves the patient for HCT)
* Patients who are positive for human immunodeficiency virus (HIV)
* Females who are pregnant or breast-feeding
* Fertile men or women who are unwilling to use contraceptives during HCT and up to 12 months post-treatment
* Patients with fungal pneumonia with radiological progression after receipt of amphotericin formulation or mold-active azoles for greater than 1 month will not be eligible for this protocol (either regimen A or B)
* Donors: Identical twin
* Donors: Pregnancy
* Donors: HIV positive
* Donors: A positive anti-donor cytotoxic cross match is absolute donor exclusion
* Donors: If a patient is homozygous at a particular loci, mismatching at that loci is not allowed due to an isolated graft rejection vector, i.e., patient A*0101 and the donor is A*0101, A*0201; such a mismatch may increase the risk of graft rejection; if patient and donor pairs are both homozygous at a mismatched loci, they are considered a two-HLA antigen mismatch, i.e., the patient is A*0101 and the donor is A*0201, and this type of mismatch is not allowed
* Donor: Donor < 6 months old, > 75 years old

Max Age: 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2006-06; Primary Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauri Burroughs, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (6):
- United States (6):
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Chemotherapy, Low Dose Radiation): CONDITIONING REGIMEN: *Patients with no life-threatening viral or fungal infections within 1 month before the planned HCT receive alemtuzumab IV over 6 hours on day -10 and fludarabine phosphate IV over 30 minutes on days -4 to -2. They also undergo low-dose TBI on day 0. Patients with HLH, IPEX syndrome, DiGeorge syndrome, or life-threatening viral or fungal infections within 1 month before the planned HCT receive fludarabine phosphate IV over 30 minutes on days -4 to -2 and undergo 2 low doses of TBI on day 0.
  HEMATOPOIETIC CELL TRANSPLANTATION: Patients undergo HCT on day 0. IMMUNOSUPPRESSION: Patients receive cyclosporine IV or PO 2-3 times daily beginning on day -3 and continuing until day 100 followed by a taper until day 180. They also receive mycophenolate mofetil IV or PO 3 times daily beginning on day 0 and continuing until day 40 followed by a taper until day 96.
  Alemtuzumab: Given IV Allogeneic Bone Marrow Transplantation: Undergo HCT Allogeneic Hematopoiet
Period: Overall Study
Arm/Group | Treatment (Chemotherapy, Low Dose Radiation)
Started | 29
Completed | 28
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemotherapy, Low Dose Radiation)
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 22
  More than one race | 4
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Achieve Greater Than 50% Donor T-cell Chimerism
Description: The study will be considered a success and the protocol worthy of further study if there is sufficient evidence that this rate is greater than the 50% rate observed in the most recently transplanted patients with nonmalignant disorders. Analyses will be carried out separately for the alemtuzumab recipients and the TBI recipients. We will be 80% confidence of success if a one-sided 80% confidence interval for the proportion of patients with successful chimerism exceeds 50%. Cumulative incidence will be used to evaluate the probability of chimerism.
Time Frame: At 1 year post transplant
Population: Excludes 9 patients who expired prior to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, Low Dose Radiation)
Number analyzed (Participants) | 19
Participants | 13

2. Secondary Outcome: Overall Survival
Description: Number of patients alive at 1 year
Time Frame: 1 year
Population: Excludes 3 patients with graft rejection and second transplant prior to 1 year.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, Low Dose Radiation)
Number analyzed (Participants) | 25
Participants | 19

3. Secondary Outcome: Immune Reconstitution by 1 Year Post Transplant
Description: Number of patients with normal range CD3 at 1 year post transplant
Time Frame: 1 year
Population: Excludes 16 patients: 13 patients who did not achieve 1 year time point (9 expired, 4 went to second transplant) and 3 patients for whom no data was sent at 1 year from external site
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (Chemotherapy, Low Dose Radiation): CONDITIONING REGIMEN: *Patients with no life-threatening viral or fungal infections within 1 month before the planned HCT receive alemtuzumab IV over 6 hours on day -10 and fludarabine phosphate IV over 30 minutes on days -4 to -2. They also undergo low-dose TBI on day 0. Patients with HLH, IPEX syndrome, DiGeorge syndrome, or life-threatening viral or fungal infections within 1 month before the planned HCT receive fludarabine phosphate IV over 30 minutes on days -4 to -2 and undergo 2 low doses of TBI on day 0.
  HEMATOPOIETIC CELL TRANSPLANTATION: Patients undergo HCT on day 0. IMMUNOSUPPRESSION: Patients receive cyclosporine IV or PO 2-3 times daily beginning on day -3 and continuing until day 100 followed by a taper until day 180. They also receive mycophenolate mofetil IV or PO 3 times daily beginning on day 0 and continuing until day 40 followed by a taper until day 96.
  Alemtuzumab: Given IV Allogeneic Bone Marrow Transplantation: Undergo HCT Allogeneic Hematopoietic S
Arm/Group | Treatment (Chemotherapy, Low Dose Radiation)
Number analyzed (Participants) | 12
Participants | 7

4. Secondary Outcome: Disease Response by 1 Year Post Transplant
Description: Number of patients at 1 year with disease response (defined as no clinical evidence of active disease and/or sufficient level of donor chimerisms to prevent disease recurrence)
Time Frame: 1 year
Population: Excludes 9 patients who expired prior to 1 year time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, Low Dose Radiation)
Number analyzed (Participants) | 19
Participants | 15

5. Secondary Outcome: Greater Than 50% CD33+ Donor Chimerisms at 1 Year Post Transplant
Description: Number of patients who achieve greater than 50% CD33+ donor chimerisms at 1 year post transplant.
Time Frame: 1 year
Population: Excludes 9 patients who expired prior to 1 year time point
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, Low Dose Radiation)
Number analyzed (Participants) | 19
Participants | 8

6. Secondary Outcome: Greater Than 50% CD19+ Donor Chimerisms at 1 Year Post Transplant
Description: Number of Patients Who Achieve Greater Than 50% CD19+ Donor Chimerisms at 1 Year Post Transplant
Time Frame: 1 year
Population: Excludes 9 patients who expired prior to 1 year time point
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (Chemotherapy, Low Dose Radiation): CONDITIONING REGIMEN: *Patients with no life-threatening viral or fungal infections within 1 month before the planned HCT receive alemtuzumab IV over 6 hours on day -10 and fludarabine phosphate IV over 30 minutes on days -4 to -2. They also undergo low-dose TBI on day 0. Patients with HLH, IPEX syndrome, DiGeorge syndrome, or life-threatening viral or fungal infections within 1 month before the planned HCT receive fludarabine phosphate IV over 30 minutes on days -4 to -2 and undergo 2 low doses of TBI on day 0.
  HEMATOPOIETIC CELL TRANSPLANTATION: Patients undergo HCT on day 0.
  IMMUNOSUPPRESSION: Patients receive cyclosporine IV or PO 2-3 times daily beginning on day -3 and continuing until day 100 followed by a taper until day 180. They also receive mycophenolate mofetil IV or PO 3 times daily beginning on day 0 and continuing until day 40 followed by a taper until day 96.
  Alemtuzumab: Given IV Allogeneic Bone Marrow Transplantation: Undergo HCT Allogeneic Hematopoietic
Arm/Group | Treatment (Chemotherapy, Low Dose Radiation)
Number analyzed (Participants) | 19
Participants | 16

7. Secondary Outcome: Clinical Significant Infection, Requiring Treatment, Within 100 Days Post Transplant
Description: Number of patients who experienced a clinical significant infection, requiring treatment, within 100 days post transplant.
Time Frame: 100 days
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (Chemotherapy, Low Dose Radiation): CONDITIONING REGIMEN: *Patients with no life-threatening viral or fungal infections within 1 month before the planned HCT receive alemtuzumab IV over 6 hours on day -10 and fludarabine phosphate IV over 30 minutes on days -4 to -2. They also undergo low-dose TBI on day 0. Patients with HLH, IPEX syndrome, DiGeorge syndrome, or life-threatening viral or fungal infections within 1 month before the planned HCT receive fludarabine phosphate IV over 30 minutes on days -4 to -2 and undergo 2 low doses of TBI on day 0.
  HEMATOPOIETIC CELL TRANSPLANTATION: Patients undergo HCT on day 0. IMMUNOSUPPRESSION: Patients receive cyclosporine IV or PO 2-3 times daily beginning on day -3 and continuing until day 100 followed by a taper until day 180. They also receive mycophenolate mofetil IV or PO 3 times daily beginning on day 0 and continuing until day 40 followed by a taper until day 96.
  Alemtuzumab: Given IV Allogeneic Bone Marrow Transplantation: Undergo HCT Allogeneic Hematopoietic Ste
Arm/Group | Treatment (Chemotherapy, Low Dose Radiation)
Number analyzed (Participants) | 28
Participants | 21

8. Secondary Outcome: Number of Patients Diagnosed With Acute GVHD
Description: Number of patients diagnosed with acute GVHD by Day 100 post transplant
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, Low Dose Radiation)
Number analyzed (Participants) | 28
Participants | 18

9. Secondary Outcome: Number of Patients Diagnosed With Overall Grade 1 or Grade 2 Acute GVHD
Description: Number of patients diagnosed with overall grade I or grade II acute GVHD by Day 100 post transplant
Time Frame: Day 100
Population: Excludes 10 patients who were not diagnosed with acute GVHD
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, Low Dose Radiation)
Number analyzed (Participants) | 18
Participants | 12

10. Secondary Outcome: Number of Patients Diagnosed With Overall Grade III or Grade IV Acute GVHD
Description: Number of patients diagnosed with overall Grade III or Grade IV Acute GVHD by Day 100 post transplant
Time Frame: Day 100
Population: Excludes 10 patients who were not diagnosed with acute GVHD
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, Low Dose Radiation)
Number analyzed (Participants) | 18
Participants | 6

11. Secondary Outcome: Number of Patients Diagnosed With Chronic GVHD
Description: Number of patients diagnosed with chronic GVHD within 1 year post transplant
Time Frame: 1 year
Population: Excludes 6 patients who expired prior to Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, Low Dose Radiation)
Number analyzed (Participants) | 22
Participants | 8

ADVERSE EVENTS:
Time Frame: Day 200 post initiation of conditioning therapy
Arm/Group | Treatment (Chemotherapy, Low Dose Radiation)
All-Cause Mortality (participants affected / at risk) | 9/28
Serious Adverse Events (participants affected / at risk) | 10/28
Other Adverse Events (participants affected / at risk) | 13/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy, Low Dose Radiation) (N=28)
Pericardial Effusion (Cardiac disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperbilirubinemia (Hepatobiliary disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Cardiorspiratory Failure (Cardiac disorders) | 3 (3)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy, Low Dose Radiation) (N=28)
Hyperbilirubinemia (Hepatobiliary disorders) | 6 (7)
Hypertension (Cardiac disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fever of Unknown Origin (Infections and infestations) | 3 (3)
Tachycardia (Cardiac disorders) | 1 (1)
Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal Insufficiency (Renal and urinary disorders) | 1 (1)
Renal Failure, requiring dialysis (Renal and urinary disorders) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Cardiovascular, not otherwise specified (Cardiac disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bleeding - Vaginal (Blood and lymphatic system disorders) | 1 (2)
Bleeding - Lung (Blood and lymphatic system disorders) | 1 (1)
Bleeding - GI (Blood and lymphatic system disorders) | 1 (1)
Bleeding - CNS (Blood and lymphatic system disorders) | 1 (1)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No